CLINICAL TRIAL: NCT03703791
Title: Peanut Allergy Oral Immunotherapy Study of AR101 for Desensitization in Children and Adolescents: Real World, Open Label, Quality of Life Study
Brief Title: Real World, Open Label, QOL Assessment of Peanut Immunotherapy AR101 in Children and Adolescents
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor terminated study; no impact on overall benefit risk evaluation of AR101
Sponsor: Aimmune Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARC009; 2018-000326-58 (EudraCT Number)
Record Dates: First submitted 2018-10-09; First posted 2018-10-12 (Actual); Results first posted 2021-07-13 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-06

CONDITIONS: Peanut Allergy
Keywords: AR101; Characterized Peanut Allergen (CPNA); (Characterized Peanut Allergen) OIT; Peanut Allergy; Allergy; Peanut-Allergic Children; Peanut-Allergic Adolescents; Desensitization; Quality of Life; OIT (oral immunotherapy); CODIT (TM) Characterized Oral Desensitization Immunotherapy (TM)
MeSH Terms: conditions — Peanut Hypersensitivity; Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1 (AR101 Treatment + standard of care) (Active Comparator): Subjects receiving AR101 treatment will have 3 consecutive AR101 dosing periods before exiting (completing) the study: initial dose escalation, up dosing, and maintenance.
  Interventions: Biological: AR101
- Group 2 (Standard of Care Treatment) (No Intervention): Subjects receiving standard of care alone will have approximately 18 months of observation before study exit, with an OLFC (open label food challenge) approximately 12 months after randomization.

INTERVENTIONS:
Biological: AR101 — AR101 powder
  Arms: Group 1 (AR101 Treatment + standard of care)

SUMMARY:
To compare the HRQOL of AR101 characterized oral desensitization immunotherapy (CODIT™) in combination with standard of care (peanut avoidance, education) versus standard of care alone in peanut-allergic subjects aged 4 to 17 years.

DETAILED DESCRIPTION:
This is a phase 3b, randomized, open label, European study of the HRQOL of AR101 in combination with standard of care compared with standard of care alone in approximately 200 peanut-allergic subjects aged 4 to 17 years, inclusive.

ELIGIBILITY:
Key Inclusion Criteria:

* Age 4 through 17 years
* History of physician diagnosed IgE mediated peanut allergy with characteristic signs and symptoms
* Positive SPT for peanut
* Positive serum IgE to peanut
* Written informed consent from the subject's parent/guardian
* Written assent from the subject as appropriate
* Use of effective birth control by sexually active female subjects of childbearing potential

Key Exclusion Criteria:

* Uncertain clinical diagnosis of peanut allergy
* History of severe or life threatening episode of anaphylaxis or anaphylactic shock within 60 days of screening
* Severe persistent asthma or uncontrolled mild or moderate asthma
* History of eosinophilic esophagitis, other eosinophilic gastrointestinal disease, severe gastroesophageal reflux disease, symptoms of dysphagia or recurrent gastrointestinal symptoms of undiagnosed etiology
* History of a mast cell disorder, including mastocytosis, urticarial pigmentosa, and hereditary or idiopathic angioedema
* History of cardiovascular disease, including uncontrolled or inadequately controlled hypertension
* History of chronic disease (other than asthma, atopic dermatitis, or allergic rhinitis) that is, or is at significant risk of becoming, unstable or requiring a change in chronic therapeutic regimen

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2018-11-23 (Actual); Study Completion 2018-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Director of Regulatory Affairs, Study Director — Aimmune Therapeutics
Locations (11):
- Spain (11):
  - Hospital Universitario Germans Trias i Pujol, Badalona, Barcelona
  - Corporacio Sanitaria Parc Tauli, Sabadell, Barcelona
  - Hospital Universitario Severo Ochoa, Leganés, Madrid
  - Hospital Universitario Vall d'Hebron - PPDS, Barcelona
  - Hospital Infantil Universitario Niño Jesus, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Complejo Hospitalario de Navarra, Pamplona
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Three subjects were screened, 1 subject was randomly assigned to standard of care alone.
Groups:
- Group 1 (AR101 Treatment + Standard of Care): Subjects receiving AR101 treatment will have 3 consecutive AR101 dosing periods before exiting (completing) the study: initial dose escalation, up dosing, and maintenance, with an OLFC (open label food challenge) approximately 12 months after randomization.
  AR101: AR101 powder
Period: Overall Study
Arm/Group | Group 1 (AR101 Treatment + Standard of Care) | Group 2 (Standard of Care Treatment)
Started | 0 | 1
Completed | 0 | 0
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Population: The study was terminated early based on the sponsor's conclusion that HRQOL data relevant to peanut allergy could be generated by alternative means.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 (AR101 Treatment + Standard of Care) | Group 2 (Standard of Care Treatment) | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Customized [Count of Participants; unit: Participants]
  14 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Health-related Quality of Life
Description: The primary analyses will use scores from a family of proxy- and self-reported disease-specific HRQOL measures to assess the HRQOL of peanut-allergic subjects treated with AR101 or standard of care alone during the study. The relevant disease-specific HRQOL questionnaires include the FAQLQ-PF (parent form), FAQLQ-PFT (parent form teenager), FAQLQ-CF (child form), FAQLQ-TF (teenager form), FAIM-PF (parent form), FAIM-PFT (parent form teenager), FAIM-CF (child form), and FAIM-TF (teenager form).
Time Frame: 18 months per subject, approximately 30 months for the study
Population: No HRQOL, efficacy, or safety measurements were collected due to the sponsor's decision to terminate the study early.
Groups:
- Group 1 (AR101 Treatment + Standard of Care): Subjects receiving AR101 treatment will have 3 consecutive AR101 dosing periods before exiting (completing) the study: initial dose escalation, up dosing, and maintenance with an OLFC (open label food challenge) approximately 12 months after randomization.
  AR101: AR101 powder
Arm/Group | Group 1 (AR101 Treatment + Standard of Care) | Group 2 (Standard of Care Treatment)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: No HRQOL, efficacy, or safety assessments were performed due to the sponsor's decision to terminate the study early.
Description: No HRQOL, efficacy, or safety assessments were performed due to the sponsor's decision to terminate the study early.
Arm/Group | Group 1 (AR101 Treatment + Standard of Care) | Group 2 (Standard of Care Treatment)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
* Institutions cannot publish until the multi-center sponsor publication is published
* Or, institutions cannot publish until 18 months after study completion
* And Sponsor review of any publications is required prior to any institution publications according to contractual agreements

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-11): https://cdn.clinicaltrials.gov/large-docs/91/NCT03703791/Prot_SAP_001.pdf